CLINICAL TRIAL: NCT01721772
Title: A Phase 3, Randomized, Double-Blind Study of BMS-936558 vs Dacarbazine in Subjects With Previously Untreated, Unresectable or Metastatic Melanoma
Brief Title: Study of Nivolumab (BMS-936558) Compared With Dacarbazine in Untreated, Unresectable, or Metastatic Melanoma
Acronym: CheckMate 066
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA209-066; 2012-003718-16 (EudraCT Number)
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Results first posted 2016-02-25 (Estimated); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Dacarbazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab, 3 mg/kg (Experimental): Participants received nivolumab, 3 mg/kg, solution administered Intravenously (IV) every 2 weeks until disease progression, discontinuation due to toxicity, withdrawal of consent, or study completion. Eligible participants may switch to nivolumab at 480mg every 4 weeks until documented disease progression, discontinuation, withdrawal of consent or the study ends.
  Interventions: Biological: BMS-936558 (Nivolumab); Drug: Placebo matching Dacarbazine
- Dacarbazine, 1000 mg/m^2 (Active Comparator): Participants received dacarbazine, 1000 mg/m^2, solution administered IV every 3 weeks until disease progression, discontinuation due to toxicity, withdrawal of consent, or study completion. Eligible participants may cross-over to nivolumab open label treatment, either 3 mg/kg every 2 weeks or 480mg every 4 weeks until documented disease progression, discontinuation, withdrawal of consent or the study ends.
  Interventions: Biological: Placebo matching BMS-936558 (Nivolumab); Drug: Dacarbazine

INTERVENTIONS:
Biological: BMS-936558 (Nivolumab)
  Arms: Nivolumab, 3 mg/kg
Biological: Placebo matching BMS-936558 (Nivolumab)
  Arms: Dacarbazine, 1000 mg/m^2
Drug: Dacarbazine
  Arms: Dacarbazine, 1000 mg/m^2
Drug: Placebo matching Dacarbazine
  Arms: Nivolumab, 3 mg/kg

SUMMARY:
The purpose of this study is to compare the clinical benefit, as measured by overall survival, of nivolumab with that of. dacarbazine in patients with previously untreated, unresectable, or metastatic melanoma

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Men and women ≥18 years of age
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Untreated and histologically confirmed unresectable Stage III or Stage IV melanoma, as per the staging system of the American Joint Committee on Cancer
* Measurable disease as per Response Evaluation Criteria in Solid Tumors 1.1
* Tumor tissue from an unresectable or metastatic site of disease must be provided for biomarker analyses
* Known BRAF wild-type, as per regionally acceptable V600 mutational status testing. BRAF mutant patients and those with indeterminate or unknown BRAF status are not permitted to randomize

Exclusion Criteria:

* Active brain metastases or leptomeningeal metastases
* Ocular melanoma
* Any active, known, or suspected autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2013-01-18 (Actual); Primary Completion 2014-06-24 (Actual); Study Completion 2021-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (73):
- Argentina (3):
  - Fundacion Cidea, Buenos Aires, Distrito Federal
  - Instituto Medico Especialazado Alexander Fleming, Buenos Aires
  - Instituto Oncologico De Cordoba, Córdoba
- Australia (9):
  - Local Institution, Camperdown, New South Wales
  - Coffs Harbour Health Campus, Coffs Harbour, New South Wales
  - Local Institution - 0006, North Sydney, New South Wales
  - Local Institution, Westmead, New South Wales
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Local Institution, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Cabrini Hospital, Malvern, Victoria
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Local Institution - 0039, Vancouver, British Columbia
  - Qe Ii Health Science Centre, Halfax, Nova Scotia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Local Institution - 0040, Montreal, Quebec
- Chile (3):
  - Local Institution, Viña del Mar, Región de Valparaíso
  - Local Institution, Santiago, Santiago Metropolitan
  - Local Institution, Santiago
- Denmark (3):
  - Aarhus Universitetshospital, Aarhus
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense
- Local Institution - 0035, Helsinki, Finland
- France (6):
  - Hopital Saint Andre, Bordeaux
  - Chu Grenoble - Hopital Albert Michallon, Grenoble
  - Chru De Lille - Hopital Claude Huriez, Lille
  - Hopital St Eloi, Montpellier
  - Hopital Saint Louis, Paris
  - Local Institution - 0013, Villejuif
- Germany (12):
  - Local Institution, Würzburg, Bavaria
  - Local Institution, Cologne
  - Local Institution, Essen
  - Local Institution, Gera
  - Local Institution, Göttingen
  - Local Institution, Heidelberg
  - Local Institution, Kiel
  - Local Institution, Magdeburg
  - Local Institution, Mainz
  - Local Institution, Nuremberg
  - Local Institution, Recklinghausen
  - Local Institution, Tübingen
- Greece (2):
  - Laiko Hospital, Athens
  - Metropolitan Hospital, Neo Faliro
- Israel (3):
  - Local Institution, Haifa
  - Local Institution, Jerusalem
  - Local Institution, Tel Litwinsky
- Italy (9):
  - Local Institution, Bari
  - Local Institution, Bergamo
  - Local Institution, Genova
  - Local Institution, Meldola (fc)
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Padua
  - Local Institution, Roma
  - Local Institution, Siena
- Mexico (4):
  - Local Institution, Leon, Guanajato, Guanajuato
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Tlalpan, Mexico City
  - Local Institution, Morelia, Michoacán
- Local Institution, Oslo, Norway
- Poland (3):
  - Local Institution, Gdansk
  - Local Institution, Lodz
  - Local Institution, Warsaw
- Spain (5):
  - Local Institution, Donostia / San Sebastian, Guipuzcoa
  - Local Institution - 0056, Barcelona
  - Local Institution, Madrid
  - Local Institution, Seville
  - Local Institution, Valencia
- Sweden (3):
  - Local Institution, Gothenberg
  - Local Institution, Lund
  - Local Institution, Umeå

REFERENCES:
- [Derived] Long GV, Larkin J, Schadendorf D, Grob JJ, Lao CD, Marquez-Rodas I, Wagstaff J, Lebbe C, Pigozzo J, Robert C, Ascierto PA, Atkinson V, Postow MA, Atkins MB, Sznol M, Callahan MK, Topalian SL, Sosman JA, Kotapati S, Thakkar PK, Ritchings C, Pe Benito M, Re S, Soleymani S, Hodi FS. Pooled Long-Term Outcomes With Nivolumab Plus Ipilimumab or Nivolumab Alone in Patients With Advanced Melanoma. J Clin Oncol. 2025 Mar 10;43(8):938-948. doi: 10.1200/JCO.24.00400. Epub 2024 Nov 6. PMID 39504507
- [Derived] Robert C, Long GV, Brady B, Dutriaux C, Di Giacomo AM, Mortier L, Rutkowski P, Hassel JC, McNeil CM, Kalinka EA, Lebbe C, Charles J, Hernberg MM, Savage KJ, Chiarion-Sileni V, Mihalcioiu C, Mauch C, Arance A, Cognetti F, Ny L, Schmidt H, Schadendorf D, Gogas H, Zoco J, Re S, Ascierto PA, Atkinson V. Five-Year Outcomes With Nivolumab in Patients With Wild-Type BRAF Advanced Melanoma. J Clin Oncol. 2020 Nov 20;38(33):3937-3946. doi: 10.1200/JCO.20.00995. Epub 2020 Sep 30. PMID 32997575
- [Derived] Ascierto PA, Long GV, Robert C, Brady B, Dutriaux C, Di Giacomo AM, Mortier L, Hassel JC, Rutkowski P, McNeil C, Kalinka-Warzocha E, Savage KJ, Hernberg MM, Lebbe C, Charles J, Mihalcioiu C, Chiarion-Sileni V, Mauch C, Cognetti F, Ny L, Arance A, Svane IM, Schadendorf D, Gogas H, Saci A, Jiang J, Rizzo J, Atkinson V. Survival Outcomes in Patients With Previously Untreated BRAF Wild-Type Advanced Melanoma Treated With Nivolumab Therapy: Three-Year Follow-up of a Randomized Phase 3 Trial. JAMA Oncol. 2019 Feb 1;5(2):187-194. doi: 10.1001/jamaoncol.2018.4514. PMID 30422243
- [Derived] Long GV, Tykodi SS, Schneider JG, Garbe C, Gravis G, Rashford M, Agrawal S, Grigoryeva E, Bello A, Roy A, Rollin L, Zhao X. Assessment of nivolumab exposure and clinical safety of 480 mg every 4 weeks flat-dosing schedule in patients with cancer. Ann Oncol. 2018 Nov 1;29(11):2208-2213. doi: 10.1093/annonc/mdy408. PMID 30215677
- [Derived] Long GV, Weber JS, Larkin J, Atkinson V, Grob JJ, Schadendorf D, Dummer R, Robert C, Marquez-Rodas I, McNeil C, Schmidt H, Briscoe K, Baurain JF, Hodi FS, Wolchok JD. Nivolumab for Patients With Advanced Melanoma Treated Beyond Progression: Analysis of 2 Phase 3 Clinical Trials. JAMA Oncol. 2017 Nov 1;3(11):1511-1519. doi: 10.1001/jamaoncol.2017.1588. PMID 28662232
- [Derived] Robert C, Long GV, Brady B, Dutriaux C, Maio M, Mortier L, Hassel JC, Rutkowski P, McNeil C, Kalinka-Warzocha E, Savage KJ, Hernberg MM, Lebbe C, Charles J, Mihalcioiu C, Chiarion-Sileni V, Mauch C, Cognetti F, Arance A, Schmidt H, Schadendorf D, Gogas H, Lundgren-Eriksson L, Horak C, Sharkey B, Waxman IM, Atkinson V, Ascierto PA. Nivolumab in previously untreated melanoma without BRAF mutation. N Engl J Med. 2015 Jan 22;372(4):320-30. doi: 10.1056/NEJMoa1412082. Epub 2014 Nov 16. PMID 25399552
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 418 were randomized (210 to nivolumab, 208 to dacarbazine) and 411 received treatment (206 with nivolumab, 205 with dacarbazine).
Groups:
- Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine: Participants received nivolumab, 3 mg/kg, solution administered Intravenously (IV) every 2 weeks with placebo-matching dacarbazine solution administered IV every 3 weeks, until disease progression, discontinuation due to toxicity, withdrawal of consent, or study completion
- Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab: Participants received dacarbazine 1000 mg/m^2, solution administered IV every 3 weeks with placebo-matching nivolumab solution administered IV every 2 weeks until disease progression, discontinuation due to toxicity, withdrawal of consent, or study completion
Period: Pre-Treatment
Arm/Group | Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine | Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab
Started (Randomized) | 210 | 208
Completed (Moving to the treatment period) | 206 | 205
Not Completed | 4 | 3
Not completed — Participant no longer meets study criteria | 3 | 1
Not completed — Poor/non-compliance | 0 | 1
Not completed — Participant withdrew consent | 0 | 1
Not completed — Adverse event unrelated to study drug | 1 | 0
Period: Treatment
Arm/Group | Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine | Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab
Started (Treated) | 206 | 205
Completed | 0 | 0
Not Completed | 206 | 205
Not completed — Disease progression | 119 | 168
Not completed — Study drug toxicity | 19 | 10
Not completed — Adverse event unrelated to study drug | 7 | 7
Not completed — Maximum clinical benefit | 16 | 4
Not completed — Other | 19 | 2
Not completed — Participant withdrew consent | 2 | 5
Not completed — Participant request to discontinue study treatment | 21 | 8
Not completed — Death | 1 | 0
Not completed — Not reported | 1 | 0
Not completed — Poor/non-compliance | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants randomized to receive treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine | Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab | Total
Number analyzed (Participants) | 210 | 208 | 418
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.6 (13.00) | 63.7 (12.60) | 62.7 (12.83)
Age, Customized [Count of Participants; unit: Participants]
  Younger than 65 years | 105 | 94 | 199
  65 to younger than 75 years | 78 | 74 | 152
  75 years and older | 27 | 40 | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 83 | 172
  Male | 121 | 125 | 246
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 209 | 207 | 416
  Black or African American | 0 | 0 | 0
  Asian | 0 | 1 | 1
  American Indian or Alaskan native | 0 | 0 | 0
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time between the date of randomization and the date of death or the last date the participant was known to be alive.
Time Frame: From date of randomization to date of death. For those without documentation of death, to the last date the participant was known to be alive, assessed up to 17 months.
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine | Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab
Number analyzed (Participants) | 210 | 208
Months | NA [NA to NA] — NA due to insufficient number of events | 10.84 [9.33 to 12.09]
Statistical Analysis 1: Comparison: Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine vs Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab; Test type: Superiority or Other; p < 0.0001, Stratified Log Rank Test; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.30 to 0.60]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Investigator-assessed PFS is defined as the time from randomization to the date of the first documented progression, as determined by the investigator, or death due to any cause, whichever occurs first. Patients who died without progressing were considered to have progressed on the date of their death. Those who did not progress or die were documented on the date of their last evaluable tumor assessment. Patients who did not have any on-study tumor assessments and did not die were documented on their date of randomization. Those who started any subsequent anticancer therapy without a prior reported progression were documented on the date of their last evaluable tumor assessment prior to initiation of subsequent anticancer therapy.
Time Frame: From date of randomization up to date of disease progression or death, up to approximately 84 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine | Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab
Number analyzed (Participants) | 210 | 208
Months | 5.06 [3.52 to 12.16] | 2.17 [2.10 to 2.50]
Statistical Analysis 1: Comparison: Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine vs Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab; Test type: Superiority or Other; p < 0.0001, Stratified Log Rank Test; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.34 to 0.56]

3. Secondary Outcome: Progression-free Survival (PFS) Rate
Description: The PFS rate at a time point is the estimated percentage of patients who have not progressed and are alive at that time point following randomization and is estimated using the Kaplan-Meier methodology.
Time Frame: From randomization to the specified timepoints, up to 84 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine | Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab
Number analyzed (Participants) | 210 | 208
Percentage of participants
  At 6 months | 48.2 [41.0 to 55.0] | 20.0 [14.6 to 26.1]
  At 12 months | 43.3 [36.3 to 50.2] | 7.4 [3.9 to 12.4]
  At 18 months | 40.5 [33.5 to 47.4] | 5.2 [2.2 to 10.2]
  At 24 months | 35.8 [29.0 to 42.6] | 5.2 [2.2 to 10.2]
  At 36 months | 32.8 [26.1 to 39.6] | 3.9 [1.3 to 8.9]
  At 48 months | 29.7 [23.2 to 36.5] | 3.9 [1.3 to 8.9]
  At 60 months | 28.4 [22.0 to 35.2] | 3.9 [1.3 to 8.9]
  At 72 months | 27.8 [21.4 to 34.5] | 3.9 [1.3 to 8.9]
  At 84 months | 25.9 [19.5 to 32.7] | 3.9 [1.3 to 8.9]

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a best overall response of Response Evaluation Criteria in Solid Tumors (RECIST) defined complete response (CR) or partial response (PR). RECIST, volume 1.1 for target lesions: CR=disappearance of all target lesions; PR=at least a 30% decrease in the sum of the longest dimension (LD) of target lesions, taking as reference the baseline sum LD; stable disease=neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum LD since the treatment started; PD=at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions, and the sum LD must have an absolute increase of ≥5 mm.
Time Frame: Tumor assessments beginning at 9 weeks following randomization and continuing every 6 weeks for the first year, then every 12 weeks thereafter until disease progression or death, assessed to 94 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine | Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab
Number analyzed (Participants) | 210 | 208
Percentage of participants | 42.4 [35.6 to 49.4] | 14.4 [9.9 to 19.9]
Statistical Analysis 1: Comparison: Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine vs Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.43, 95% CI 2-sided [2.75 to 7.13]

5. Secondary Outcome: Overall Survival by Programmed Cell Death Ligand 1 (PD-L1) Expression Level
Description: Overall Survival is defined as the time between the date of randomization and the date of death or the last date the participant was known to be alive. PD-L1 expression level is defined as the percent of tumor cells demonstrating plasma membrane PD-L1-staining in a minimum of 100 evaluable tumor cells per a Dako PD-L1 IHC (immunohistochemistry) assay (referred to as quantifiable PD-L1 expression). Assessment of OS by PD-L1 expression as measured by a validated assay and comparing OS in patients with tumor PD-L1 expression ≥5% (PD-L1 positive) versus patients with tumor PD-L1 expression <5% (PD-L1 negative). Tumor tissue samples for PD-L1 testing were collected at screening from metastatic or unresectable sites prior to randomization.
Time Frame: From date of randomization to date of disease progression or death, up to approximately 94 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine | Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab
Number analyzed (Participants) | 210 | 208
Months
  PD-L1 positive participants (cutoff=5%): number analyzed (Participants) | 74 | 74
  PD-L1 positive participants (cutoff=5%) | 53.36 [31.47 to NA] — Upper limit not reached due to insufficient number of events | 12.39 [9.33 to 18.99]
  PD-L1 negative/indeterminate participants (cutoff=5%): number analyzed (Participants) | 136 | 134
  PD-L1 negative/indeterminate participants (cutoff=5%) | 26.97 [16.36 to 39.79] | 10.84 [8.38 to 12.25]
Statistical Analysis 1: Comparison: Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine vs Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab; Test type: Superiority or Other; Unstratified Hazard Ratio = 0.37, 95% CI 2-sided [0.24 to 0.56] — PD-L1 positive group
Statistical Analysis 2: Comparison: Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine vs Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab; Test type: Superiority or Other; Unstratified Hazard Ratio = 0.60, 95% CI 2-sided [0.45 to 0.80] — PD-L1 negative group

6. Primary Outcome: Overall Survival (OS) Rate
Description: OS rate is calculated as the percentage of participants alive at the indicated timepoints
Time Frame: From randomization to 6 months and or to 12 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine | Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab
Number analyzed (Participants) | 210 | 208
Percentage of participants
  At 6 months | 84.1 [78.3 to 88.5] | 71.8 [64.9 to 77.6]
  At 12 months | 72.9 [65.5 to 78.9] | 42.1 [33.0 to 50.9]

7. Secondary Outcome: Change From Baseline in Health-related Quality of Life (HRQoL) Scores
Description: HRQoL is evaluated by mean changes from baseline in the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) global health status/quality of life composite scale in all randomized patients. The QLQ-30 is a cancer-specific, self-administered questionnaire that contains 30 questions, covering global, functional, and symptom scales. Scores range from 0 to 100. Higher scores on global and functional scales indicate better quality of life (QoL), while higher scores on the symptom scales indicate declining QoL.
Time Frame: At baseline and every 6 weeks for 12 months and at follow-up visits 1 and 2, assessed up to 93 months
Population: All randomized participants with available measurements
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine | Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab
Number analyzed (Participants) | 210 | 208
Units on a scale
  Week 7: number analyzed (Participants) | 126 | 115
  Week 7 | 1.39 (19.46) | 2.32 (20.52)
  Week 13: number analyzed (Participants) | 95 | 59
  Week 13 | 1.49 (18.91) | 3.81 (16.33)
  Week 19: number analyzed (Participants) | 87 | 37
  Week 19 | 3.07 (16.58) | 3.15 (17.16)
  Week 25: number analyzed (Participants) | 71 | 33
  Week 25 | 3.52 (20.25) | -0.76 (21.28)
  Week 31: number analyzed (Participants) | 66 | 20
  Week 31 | 2.53 (20.46) | 4.17 (17.83)
  Week 37: number analyzed (Participants) | 64 | 14
  Week 37 | 3.26 (17.61) | 7.14 (18.45)
  Week 43: number analyzed (Participants) | 69 | 8
  Week 43 | 1.69 (20.24) | -1.04 (18.06)
  Week 49: number analyzed (Participants) | 60 | 5
  Week 49 | 4.31 (18.95) | 3.33 (13.94)
  Week 55: number analyzed (Participants) | 57 | 6
  Week 55 | 2.92 (18.26) | 12.50 (23.42)
  Week 61: number analyzed (Participants) | 56 | 3
  Week 61 | 1.79 (18.72) | 13.89 (17.35)
  Week 67: number analyzed (Participants) | 56 | 2
  Week 67 | 2.08 (21.92) | 8.33 (11.79)
  Week 73: number analyzed (Participants) | 48 | 2
  Week 73 | 4.69 (17.10) | 12.50 (5.89)
  Week 79: number analyzed (Participants) | 46 | 2
  Week 79 | 5.62 (18.84) | 8.33 (11.79)
  Week 85: number analyzed (Participants) | 41 | 2
  Week 85 | 3.05 (19.43) | 12.50 (5.89)
  Week 91: number analyzed (Participants) | 41 | 2
  Week 91 | 3.66 (20.92) | 16.67 (0.00)
  Week 97: number analyzed (Participants) | 39 | 2
  Week 97 | 4.27 (19.48) | 8.33 (11.79)
  Week 103: number analyzed (Participants) | 39 | 1
  Week 103 | 6.20 (19.56) | 0.00 (0.00)
  Week 109: number analyzed (Participants) | 37 | 2
  Week 109 | 3.83 (20.75) | 8.33 (11.79)
  Week 115: number analyzed (Participants) | 34 | 1
  Week 115 | 4.17 (21.15) | 0.00 (0.00)
  Week 121: number analyzed (Participants) | 34 | 1
  Week 121 | 1.47 (20.25) | 0.00 (0.00)
  Week 127: number analyzed (Participants) | 32 | 0
  Week 127 | -0.26 (19.91) |
  Week 133: number analyzed (Participants) | 29 | 1
  Week 133 | 3.16 (22.09) | 16.67 (NA) — Insufficient number of participants to calculate standard deviation
  Week 139: number analyzed (Participants) | 30 | 1
  Week 139 | 1.11 (21.86) | 16.67 (NA) — Insufficient number of participants to calculate standard deviation
  Week 145: number analyzed (Participants) | 32 | 1
  Week 145 | 4.69 (20.07) | 16.67 (NA) — Insufficient number of participants to calculate standard deviation
  Week 151: number analyzed (Participants) | 30 | 1
  Week 151 | 1.67 (20.34) | 16.67 (NA) — Insufficient number of participants to calculate standard deviation
  Week 157: number analyzed (Participants) | 26 | 1
  Week 157 | 3.53 (22.99) | 33.33 (NA) — Insufficient number of participants to calculate standard deviation
  Week 163: number analyzed (Participants) | 21 | 1
  Week 163 | 7.94 (20.83) | 16.67 (NA) — Insufficient number of participants to calculate standard deviation
  Week 169: number analyzed (Participants) | 20 | 1
  Week 169 | 13.33 (17.61) | 33.33 (NA) — Insufficient number of participants to calculate standard deviation
  Week 175: number analyzed (Participants) | 17 | 1
  Week 175 | 7.84 (23.66) | 50.00 (NA) — Insufficient number of participants to calculate standard deviation
  Week 181: number analyzed (Participants) | 20 | 0
  Week 181 | 5.42 (21.16) |
  Week 187: number analyzed (Participants) | 18 | 1
  Week 187 | 1.85 (22.06) | 33.33 (NA) — Insufficient number of participants to calculate standard deviation
  Week 193: number analyzed (Participants) | 20 | 1
  Week 193 | 2.50 (20.96) | 16.67 (NA) — Insufficient number of participants to calculate standard deviation
  Week 199: number analyzed (Participants) | 16 | 1
  Week 199 | 6.77 (21.13) | 33.33 (NA) — Insufficient number of participants to calculate standard deviation
  Week 205: number analyzed (Participants) | 18 | 1
  Week 205 | 0.93 (24.07) | 33.33 (NA) — Insufficient number of participants to calculate standard deviation
  Week 211: number analyzed (Participants) | 17 | 0
  Week 211 | 0.49 (18.97) |
  Week 217: number analyzed (Participants) | 21 | 1
  Week 217 | 1.19 (23.32) | 33.33 (NA) — Insufficient number of participants to calculate standard deviation
  Week 223: number analyzed (Participants) | 19 | 1
  Week 223 | 5.26 (25.49) | 33.33 (NA) — Insufficient number of participants to calculate standard deviation
  Week 229: number analyzed (Participants) | 21 | 1
  Week 229 | 5.56 (23.77) | 16.67 (NA) — Insufficient number of participants to calculate standard deviation
  Week 235: number analyzed (Participants) | 17 | 0
  Week 235 | 5.39 (24.82) |
  Week 241: number analyzed (Participants) | 18 | 0
  Week 241 | 2.78 (25.72) |
  Week 247: number analyzed (Participants) | 14 | 1
  Week 247 | 5.36 (25.45) | 16.67 (NA) — Insufficient number of participants to calculate standard deviation
  Week 253: number analyzed (Participants) | 15 | 1
  Week 253 | 3.89 (26.89) | 16.67 (NA) — Insufficient number of participants to calculate standard deviation
  Week 259: number analyzed (Participants) | 13 | 1
  Week 259 | 7.05 (24.26) | 25.00 (NA) — Insufficient number of participants to calculate standard deviation
  Week 265: number analyzed (Participants) | 14 | 1
  Week 265 | 8.93 (21.55) | 33.33 (NA) — Insufficient number of participants to calculate standard deviation
  Week 271: number analyzed (Participants) | 12 | 0
  Week 271 | 6.25 (21.94) |
  Week 277: number analyzed (Participants) | 14 | 1
  Week 277 | 4.17 (21.12) | 25.00 (NA) — Insufficient number of participants to calculate standard deviation
  Week 283: number analyzed (Participants) | 12 | 1
  Week 283 | 5.56 (21.42) | 33.33 (NA) — Insufficient number of participants to calculate standard deviation
  Week 289: number analyzed (Participants) | 14 | 1
  Week 289 | 3.57 (20.86) | 33.33 (NA) — Insufficient number of participants to calculate standard deviation
  Week 295: number analyzed (Participants) | 12 | 1
  Week 295 | 3.47 (23.15) | 16.67 (NA) — Insufficient number of participants to calculate standard deviation
  Week 301: number analyzed (Participants) | 12 | 1
  Week 301 | 2.78 (23.92) | 16.67 (NA) — Insufficient number of participants to calculate standard deviation
  Week 307: number analyzed (Participants) | 11 | 1
  Week 307 | 1.52 (24.95) | 33.33 (NA) — Insufficient number of participants to calculate standard deviation
  Week 313: number analyzed (Participants) | 10 | 0
  Week 313 | 9.17 (24.04) |
  Week 319: number analyzed (Participants) | 10 | 1
  Week 319 | 3.33 (26.70) | 33.33 (NA) — Insufficient number of participants to calculate standard deviation
  Week 325: number analyzed (Participants) | 8 | 0
  Week 325 | 9.38 (25.37) |
  Week 331: number analyzed (Participants) | 7 | 1
  Week 331 | 10.71 (27.09) | 33.33 (NA) — Insufficient number of participants to calculate standard deviation
  Week 337: number analyzed (Participants) | 7 | 0
  Week 337 | 11.90 (26.29) |
  Week 343: number analyzed (Participants) | 6 | 0
  Week 343 | 16.67 (26.35) |
  Week 349: number analyzed (Participants) | 7 | 0
  Week 349 | 9.52 (26.54) |
  Week 355: number analyzed (Participants) | 5 | 0
  Week 355 | 0 (10.21) |
  Week 361: number analyzed (Participants) | 4 | 0
  Week 361 | 20.83 (30.81) |
  Week 367: number analyzed (Participants) | 3 | 0
  Week 367 | 25.00 (36.32) |
  Week 373: number analyzed (Participants) | 3 | 0
  Week 373 | 25.00 (36.32) |
  Week 379: number analyzed (Participants) | 1 | 0
  Week 379 | 8.33 (NA) — Insufficient number of participants to calculate standard deviation |
  Week 385: number analyzed (Participants) | 1 | 0
  Week 385 | 8.33 (NA) — Insufficient number of participants to calculate standard deviation |
  Week 391: number analyzed (Participants) | 1 | 0
  Week 391 | 8.33 (NA) — Insufficient number of participants to calculate standard deviation |
  Week 397: number analyzed (Participants) | 1 | 0
  Week 397 | 8.33 (NA) — Insufficient number of participants to calculate standard deviation |
  Week 403: number analyzed (Participants) | 1 | 0
  Week 403 | 8.33 (NA) — Insufficient number of participants to calculate standard deviation |

8. Post Hoc Outcome: Overall Survival (OS) Extended
Description: OS is defined as the time between the date of randomization and the date of death. For those without documentation of death, OS will be censored on the last date the participant was known to be alive. OS data for this endpoint was collected after the primary completion date up until study completion.
Time Frame: From date of randomization to date of death. For those without documentation of death, to the last date the participant was known to be alive, assessed up to 94 months.
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine | Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab
Number analyzed (Participants) | 210 | 208
Months | 37.29 [25.40 to 51.55] | 11.17 [9.56 to 12.98]
Statistical Analysis 1: Comparison: Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine vs Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab; Test type: Superiority; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.41 to 0.65]

9. Post Hoc Outcome: Overall Survival (OS) Rate Extended
Description: OS rate is calculated as the percentage of participants alive at the indicated timepoints. Data for this endpoint was collected after the primary completion date up until study completion. The OS rate for the 6 month and 12 month timepoints reflect updated data that was collected after the primary completion date.
Time Frame: From randomization to the specified timepoints, up to 84 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine | Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab
Number analyzed (Participants) | 210 | 208
Percentage of participants
  6 months | 48.2 [41.0 to 55.0] | 20.0 [14.6 to 26.1]
  12 months | 43.3 [36.3 to 50.2] | 7.4 [3.9 to 12.4]
  18 months | 63.8 [56.8 to 70.0] | 36.7 [30.0 to 43.3]
  24 months | 57.8 [50.7 to 64.2] | 26.3 [20.4 to 32.6]
  36 months | 50.8 [43.7 to 57.5] | 21.6 [16.1 to 27.6]
  48 months | 43.8 [36.9 to 50.5] | 17.9 [12.9 to 23.6]
  60 months | 39.3 [32.6 to 46.0] | 17.4 [12.4 to 23.0]
  72 months | 37.3 [30.7 to 43.9] | 16.9 [12.0 to 22.5]
  84 months | 36.2 [29.5 to 42.8] | 16.9 [12.0 to 22.5]

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from date of randomization to study completion (up to approximately 99 months). Serious Adverse events and other adverse events were assessed from date of first dose to 100 days following date of last dose (up to approximately 97 months).
Description: All-Cause Mortality = all randomized participants SAEs and NSAEs (Other Adverse Events) = all treated participants
Arm/Group | Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine | Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab
All-Cause Mortality (participants affected / at risk) | 126/210 | 165/208
Serious Adverse Events (participants affected / at risk) | 125/206 | 119/205
Other Adverse Events (participants affected / at risk) | 191/206 | 187/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine (N=206) | Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab (N=205)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 4
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 2 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Eyelid retraction (Eye disorders) | 0 | 1
Retinal vein thrombosis (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Ascites (Gastrointestinal disorders) | 3 | 1
Colitis (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Enterocolitis (Gastrointestinal disorders) | 0 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric mucosal lesion (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Chills (General disorders) | 0 | 1
Death (General disorders) | 1 | 1
Fatigue (General disorders) | 2 | 3
General physical health deterioration (General disorders) | 6 | 6
Infusion site reaction (General disorders) | 0 | 1
Injection site reaction (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 2 | 6
Pyrexia (General disorders) | 4 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 3 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 0
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 3 | 2
Coronavirus infection (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 2
Infected cyst (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Infusion site infection (Infections and infestations) | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0
Blood calcium decreased (Investigations) | 0 | 1
General physical condition abnormal (Investigations) | 2 | 0
Oxygen saturation decreased (Investigations) | 0 | 1
Pancreatic enzymes abnormal (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 32 | 69
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 1
Facial paresis (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 1 | 0
Neurological decompensation (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 2 | 2
Somnolence (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 2 | 2
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Device dislocation (Product Issues) | 1 | 0
Device occlusion (Product Issues) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 4
Disorientation (Psychiatric disorders) | 1 | 0
Mania (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Haematuria (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal injury (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Sarcoid-like reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1
Embolism (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab, 3 mg/kg + Placebo-matching Dacarbazine (N=206) | Dacarbazine, 1000 mg/m^2 + Placebo-matching Nivolumab (N=205)
Anaemia (Blood and lymphatic system disorders) | 26 | 24
Neutropenia (Blood and lymphatic system disorders) | 1 | 26
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 22
Hyperthyroidism (Endocrine disorders) | 11 | 3
Hypothyroidism (Endocrine disorders) | 20 | 8
Abdominal pain (Gastrointestinal disorders) | 30 | 21
Abdominal pain upper (Gastrointestinal disorders) | 17 | 12
Constipation (Gastrointestinal disorders) | 57 | 57
Diarrhoea (Gastrointestinal disorders) | 75 | 58
Dyspepsia (Gastrointestinal disorders) | 11 | 7
Nausea (Gastrointestinal disorders) | 59 | 104
Vomiting (Gastrointestinal disorders) | 34 | 54
Asthenia (General disorders) | 43 | 38
Fatigue (General disorders) | 77 | 60
Influenza like illness (General disorders) | 13 | 4
Oedema peripheral (General disorders) | 26 | 11
Pain (General disorders) | 13 | 13
Pyrexia (General disorders) | 36 | 29
Bronchitis (Infections and infestations) | 12 | 4
Influenza (Infections and infestations) | 15 | 3
Nasopharyngitis (Infections and infestations) | 34 | 10
Rhinitis (Infections and infestations) | 12 | 3
Upper respiratory tract infection (Infections and infestations) | 20 | 13
Urinary tract infection (Infections and infestations) | 13 | 11
Alanine aminotransferase increased (Investigations) | 17 | 7
Aspartate aminotransferase increased (Investigations) | 12 | 8
Blood alkaline phosphatase increased (Investigations) | 12 | 7
Blood creatinine increased (Investigations) | 12 | 6
Gamma-glutamyltransferase increased (Investigations) | 13 | 6
Platelet count decreased (Investigations) | 0 | 11
Decreased appetite (Metabolism and nutrition disorders) | 40 | 37
Hyperglycaemia (Metabolism and nutrition disorders) | 14 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 46 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 39 | 23
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 34 | 20
Dizziness (Nervous system disorders) | 14 | 15
Headache (Nervous system disorders) | 45 | 32
Anxiety (Psychiatric disorders) | 16 | 12
Insomnia (Psychiatric disorders) | 15 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 40 | 29
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 | 25
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 4
Actinic keratosis (Skin and subcutaneous tissue disorders) | 14 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 21 | 5
Erythema (Skin and subcutaneous tissue disorders) | 29 | 7
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 5 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 64 | 40
Rash (Skin and subcutaneous tissue disorders) | 63 | 29
Vitiligo (Skin and subcutaneous tissue disorders) | 37 | 3
Hypertension (Vascular disorders) | 22 | 5
Hypotension (Vascular disorders) | 5 | 11

LIMITATIONS AND CAVEATS:
An independent data monitoring committee (DMC) found that data from a DMC-requested database lock showed clear survival benefit with nivolumab and thus recommended unblinding the study and switching patients randomized to dacarbazine to nivolumab.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.